CLINICAL TRIAL: NCT04839666
Title: Incidence of Perioperative Hypersensitivity Reactions to Propofol in Children Allergic to Egg and/or Soy
Brief Title: Hypersensitivity Reactions to Propofol in Children
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Hypersensitivity; Allergy, Egg; Soy Allergy
MeSH Terms: conditions — Hypersensitivity; Egg Hypersensitivity | interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Perioperatively propofol administration

SUMMARY:
The investigators would only include the children who received propofol (Propolipid, Fresenius Kabi, Schelle, Belgium) for sedation, the investigators would exclude the children that didn't receive propofol during the procedure.

The investigators would analyze the incidence of hypersensitivity reaction to propofol in children allergic to egg, soy or both egg and soy and to compare those with the incidence of hypersensitivity reactions in children without allergy to egg and/or to soy. Those data were retrieved following longitudinal follow-up after the intervention. Allergy tests by skin and radioallergosorbent tests were performed in all children before the gastrointestinal endoscopy under anesthesia took place, but no results were known at the time of the sedation. A patient was defined as allergic to egg and/or soy if the patient had specific S-IgE level more than the normal level set by our institution (0.35 kU/L).

The investigators would also investigate the influence of other obtained parameters in the dataset (age, ASA score, weight category, type of investigation, respiratory and neurological comorbidities, respiratory infections, GERD, other allergies) on those results with multivariate analysis.

We considered that clinical features suggesting a hypersensitivity reaction present during anaesthesia were cutaneous, respiratory or cardiovascular manifestations. Depending on the severity of the reaction, necessitating prompt hemodynamic resuscitation with the administration of epinephrine, antihistamines, inhaled beta-agonists or corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic gastrointestinal endoscopy
* monitored anesthesia
* received propofol during the procedure
* allergic to egg and/or soy if the patient had specific S-IgE level more than the normal level set by our institution (0.35 kU/L)

Exclusion Criteria:

* Procedure without administration of propofol

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who underwent a surgery in UZ Brussels between the period of 01 January 2010 until 31 August 2016.
Sampling Method: Probability Sample
Enrollment: 2299 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with a hypersensitivity reaction | minutes, during surgery
  clinical features suggesting a hypersensitivity reaction present during anaesthesia were cutaneous, respiratory or cardiovascular manifestations.

SECONDARY OUTCOMES:
Influence of gender on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of gender on hypersensitivity reaction
Influence of ASA on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of ASA on hypersensitivity reaction
Influence of type of procedure on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of type of procedure on hypersensitivity reaction
Influence of age on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of age on hypersensitivity reaction
Influence of weight on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of weight on hypersensitivity reaction
Influence of height on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of height on hypersensitivity reaction
Influence of the experience of the gastroenterologist on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of experience of gastroenterologist on hypersensitivity reaction
Influence of a respiratory comorbitidity on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of respiratory comorbidity on hypersensitivity reaction.
Influence of a neurological comorbidity on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of a neurological comorbidity on hypersensitivity reaction
Influence of reason for investigation on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of the reason for investigation on hypersensitivity reaction
Influence of a respiratory infection on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of a respiratory infection on hypersensitivity reaction.
Influence of GERD on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of GERD on hypersensitivity reaction
Influence of an allergy besides egg or soy on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of another allergy besides egg or soy on hypersensitivity reaction.
Influence of ketamine on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of ketamine on hypersensitivity reaction.
Influence of midazolam on hypersensitivity reaction | minutes, during surgery
  See if there is a link or influence of midazolam on hypersensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No